CLINICAL TRIAL: NCT01825161
Title: The Epidemiology, Process and Outcomes of Spine Oncology
Brief Title: The Epidemiology, Process and Outcomes of Spine Oncology (EPOSO)
Acronym: EPOSO
Status: Completed | Type: Observational
Sponsor: AO Foundation, AO Spine (Other)
Collaborators: Orthopaedic Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: SPN-12-002
Record Dates: First submitted 2013-03-28; First posted 2013-04-05 (Estimated); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Secondary Malignant Neoplasm of Vertebral Column

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main purpose of this study is to utilize a comprehensive, prospective clinical database to collect patient, diagnostic and treatment variables along with disease specific and generic health related quality of life (HRQOL) data on consecutively treated patients with metastatic spine tumors. The objectives are to determine the validity and reliability of the Spine Cancer Outcomes Questionnaire (SCOQ) for use in the assessment of spine tumor outcomes, to determine if the Spine Instability Neoplastic Score (SINS) Classification is a valid tool for predicting the stability of spine in metastatic spine disease, and to determine the efficacy of surgery versus radiotherapy for the treatment of impending instability secondary to metastatic disease of the spine.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age between 18 and 75 years
* Able to read and write English at an elementary level
* Diagnosis of metastatic tumor of the spine

Exclusion Criteria:

* The primary cancer site is central nervous system or spine
* History of substance abuse (recreational drugs, alcohol) within 12 months prior to screening
* Is a prisoner
* A disease or condition that would, in opinion of the investigator, preclude accurate evaluation (e.g. significant psychiatric disease)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic spine disease
Sampling Method: Non-Probability Sample
Enrollment: 454 (Actual)
Dates: Start 2013-08; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in Spine Cancer Outcomes Questionnaire (SCOQ) | 0, 6, 12, 26, 52 and 104 weeks
  This is a new questionnaire, also referred to as the Spine Oncology Self-Assessment, developed by members of the SOSG. It is made up of 5 domains: physical function, neural function, pain, mental health and social function. It was developed as a comparison to the SF-36 for patients with spine tumors. The reliability and validity of this questionnaire will be compared with the SF-36v2.

SECONDARY OUTCOMES:
Change in Pain Numeric Rating Scale (NRS) | 0, 6, 12, 26, 52 and 104 weeks
  The Pain NRS is an 11-point horizontal scale where the end points are the extremes of no pain (0) and pain as bad as it could be, or worst pain (10). It measures subjective intensity of pain and the patient rates his/her overall or average daily pain.
Change in EuroQoL 5D (EQ-5D) | 0, 6, 12, 26, 52 and 104 weeks
  The EuroQOL group developed a standardized instrument for use as a measure of health outcome. Applicable to a wide range of health conditions and treatments, it contains 5 questions and provides a simple descriptive profile and a single index value for health status. EQ-5D is designed for self-completion by respondents and is ideally suited for use in mailed surveys, in clinics and face-to-face interviews. It is cognitively simple, taking only a few minutes to complete. Instructions to respondents are included in the questionnaire.
Change in Short Form 36 version 2 (SF-36 v2) | 0, 6, 12, 26, 52 and 104 weeks
  The SF-36 v2 (Medical Outcomes Trust, Boston, MA) is a multipurpose, short-form health survey with 36 questions available in several languages. It yields an eight-scale profile of scores: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); and 8) general health perceptions. In addition, two composite scores are constructed using factorial modeling, one for physical health (Physical Composite Score - PCS) and one for mental health (Mental Composite Score - MCS).
Change in International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) | 0, 6, 12, 26, 52 and 104 weeks
  ISNCSCI is a standardized examination to determine neurologic function and has been a standard clinical assessment for patients with neurological deficit. The modified ISNCSCI used in this study will assess the Motor Score and the ASIA Impairment Scale V 1.3 only.

CONTACTS AND LOCATIONS:
Overall Officials: Charles G Fisher, MD, Principal Investigator — Vancouver General Hospital and the University of British Columbia
Locations (10):
- United States (5):
  - Kansas University Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Canada (4):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - University of Toronto Hospital, Toronto, Ontario
  - Montreal General Hospital, Montreal, Quebec
- National Center for Spinal Disorders, Budapest, Hungary

REFERENCES:
- [Derived] Barzilai O, Sahgal A, Rhines LD, Versteeg AL, Sciubba DM, Lazary A, Weber MH, Schuster JM, Boriani S, Bettegowda C, Arnold PM, Clarke MJ, Laufer I, Fehlings MG, Gokaslan ZL, Fisher CG; AO Spine Knowledge Forum Tumor. Patient-Reported and Clinical Outcomes of Surgically Treated Patients With Symptomatic Spinal Metastases: Results From Epidemiology, Process, and Outcomes of Spine Oncology (EPOSO), a Prospective, Multi-Institutional and International Study. Neurosurgery. 2024 Nov 1;95(5):1148-1157. doi: 10.1227/neu.0000000000002989. Epub 2024 Jun 4. PMID 38832791
- See also: AOSpine — http://www.aospine.org
- See also: Orthopedic Research Foundation — http://www.oref.org